CLINICAL TRIAL: NCT03987958
Title: Prospective Non-interventional Study to Describe the Effectiveness and Safety of Venetoclax in Acute Myeloid Leukemia (AML) Patients in Routine Clinical Practice (REVIVE Study)
Brief Title: A Study to Describe the Safety and Effectiveness of Venetoclax in Acute Myeloid Leukemia (AML) Patients (REVIVE Study)
Acronym: REVIVE
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-831
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia, Venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax: Participants in this observational study will receive treatment with venetoclax for AML.
  The decision to treat with venetoclax has been made independently from this observational study before participants are offered the opportunity to participate in this study.

SUMMARY:
This study will describe the safety and effectiveness of venetoclax in AML patients in routine clinical practice in Israel. The decision to treat with venetoclax is made by the physician prior to any decision regarding participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed with Acute Myeloid Leukemia (AML) and is eligible to receive venetoclax per Israel Ministry of Health.
* Participant who will be treated with venetoclax and the decision to treat with venetoclax is made by the physician prior to any decision regarding participation in this study.

Exclusion Criteria:

- Participant participating in an interventional trial within 30 days prior to starting venetoclax treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with AML treated with venetoclax in routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Time from treatment to death from any cause, up to approximately 30 months
  Overall survival is defined as the time from the date of first treatment to the date of death from any cause.

SECONDARY OUTCOMES:
Percentage of participants achieving composite complete remission (CR or CRi) | Approximately 30 months
  The percentage of participants achieving CR or CRi will be calculated based on the modified International Working Group (IWG) criteria for AML.
Time to transfusion independence | Up to 30 months
  Transfusion independence is defined as the time between date of first venetoclax treatment and absence of red blood cell (RBC) or platelet transfusion for any consecutive 8 and/or 16 week period.
Percentage of participants achieving transfusion independence | Up to 30 months
  Transfusion independence is defined as the time between date of first venetoclax treatment and absence of red blood cell (RBC) or platelet transfusion for any consecutive 8 and/or 16 week period.
Percentage of participants treated with venetoclax as compared to participants treated with other approved biologics | Up to approximately 30 months
  The percentage of participants treated with venetoclax in combination with Hypomethylating Agents (HMAs) and Low Dose Cytarabine (LDAC) will demonstrate treatment patterns of prescribing physicians.
Change in patient reported outcomes for the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire CORE (EORTC QLQ-C30) | Week 0 to approximately 30 months
  EORTC QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
Change in patient reported outcomes for the Euro Quality of Life 5 Dimensions 5 Levels Questionnaire (EQ-5D-5L) | Week 0 to approximately 30 months
  The EQ-5D-5L is a standardized, non-disease specific instrument used to measure health-related quality of life. The EQ-5D-5L assesses general health on 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The scores for the 5 dimensions are used to compute a single utility index score ranging from 0 to 1 representing the general health status of the individual, with higher scores indicating better health state.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (12):
- Israel (12):
  - Meir Medical Center /ID# 213352, Kfar Saba, Central District
  - Assuta Tel Aviv Medical Center /ID# 213371, Tel Aviv, Central District
  - HaEmek Medical Center /ID# 213370, Afula, Haifa District
  - Shaare Zedek Medical Center /ID# 228016, Jerusalem, Jerusalem
  - Hadassah /ID# 213356, Jerusalem, Jerusalem
  - ZIV Medical Center /ID# 229211, Safed, Northern District
  - Soroka University Medical Center /ID# 213369, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 213353, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 213354, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 213355, Haifa
  - Bnai Zion Medical Center /ID# 213344, Haifa
  - Rabin Medical Center. /ID# 213343, Petah Tikva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wolach O, Levi I, Nachmias B, Tavor S, Amitai I, Ofran Y, Ganzel C, Zuckerman T, Okasha D, Hellmann I, Tadmor T, Dally N, Canaani J, Stemer G, Grunspan M, Berger AJ, Frankel N, Berelovich J, Bleterman A, Barak M, Cohen R, Moshe Y. Trial eligibility, treatment patterns, and outcome for venetoclax-based therapy in AML: a prospective cohort study. Blood Adv. 2025 Apr 8;9(7):1544-1554. doi: 10.1182/bloodadvances.2024014014. PMID 39637307
- See also: Related info — https://www.rxabbvie.com/